CLINICAL TRIAL: NCT06554457
Title: Study on the Clinical Effectiveness of Oral Strong Opioids for Common Orthopedic Surgeries Following Multimodal Analgesia
Brief Title: Post Surgical Multimodal Analgesia With Oral Strong Opioids
Acronym: ORORA
Status: Not yet recruiting | Type: Observational
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Tsu-Te Yeh, Attending Surgeon, Tri-Service General Hospital
Other Study IDs: ORORA24
Record Dates: First submitted 2024-08-09; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Orthopedic Procedures; Arthroplasty; Fracture Fixation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Fracture fixation: Fracture of upper or lower limbs or pelvis requiring internal fixation surgery
  Interventions: Drug: Multimodal analgesia with oral strong opioids
- Spinal fusion: Spinal fusion surgery
  Interventions: Drug: Multimodal analgesia with oral strong opioids
- Arthroplasty: Joint replacement surgery
  Interventions: Drug: Multimodal analgesia with oral strong opioids

INTERVENTIONS:
Drug: Multimodal analgesia with oral strong opioids — Physician's choice of post-surgical multimodal analgesia with an oral strong opioid as the backbone analgesics

SUMMARY:
This is a prospective observational case study, focusing on the clinical effectiveness of oral strong opioids for pain management following common orthopedic surgeries.The study aims to evaluate the effectiveness of multimodal analgesia with oral strong opioids, reduce common opioid-related side effects, and improve patient compliance and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or older
2. Must undergo one of the following treatments:

(1) Fracture of upper or lower limbs or pelvis requiring internal fixation surgery (2) Spinal fusion surgery (3) Joint replacement surgery 3. Requiring multimodal analgesics for postoperative pain control, with oral strong opioids as the primary opioid analgesic, as assessed by his/her physician.

4. Voluntarily sign the informed consent form and agree to the collection of clinical questionnaires and medical-related information for this study.

Exclusion Criteria:

1. Patients who have not received any or have only received oral potent opioids for no more than 1 day during the postoperative hospitalization period (including those known to be intolerant or allergic to opioid medications).
2. Patients who have received or are expected to use long-acting opioid injections within 7 days before surgery or during the postoperative hospitalization period.
3. Patients who use patient-controlled analgesics for pain control after surgery.
4. Patients with a history of substance abuse or who require continuous treatment with other opioid receptor agonists or antagonists (such as naloxone or methadone).
5. Patients with a history of mental illness who continue to require medication control from 28 days before surgery and until discharge.
6. Other cases deemed ineligible by the study investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are hospitalized for the following surgical treatment may be enrolled:
  1. Fracture of upper or lower limbs or pelvis requiring internal fixation surgery
  2. Spinal fusion surgery
  3. Joint replacement surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-08-12 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in pain scores from baseline | Twice daily during hospitalization (approximately within 1 week), at the first return 1 day visit and at 3 months after surgery
  Assess the efficacy of including oral strong opioids in multimodal pain control. For this objective, we will observe changes in pain scores among participants during postoperative treatment.

SECONDARY OUTCOMES:
Occurence of adverse events | During hospitalization (approximately within 1 week)
  Avoid common adverse reactions associated with traditional morphine-like drugs, such as respiratory depression and addiction, to enhance treatment safety and patient comfort. We will monitor the occurrence rate of adverse reactions related to oral potent opioids.
Compliance of oral strong opioids | During hospitalization (approximately within 1 week)
  Improvement the convenience of analgesic medication by transitioning from injections to oral administration, making it easier for patients to accept and adhere to the treatment plan. The compliance rate of oral strong opioids will be measured.
Physician's global impression - improvement scale(CGI-I) | During hospitalization (approximately within 1 week), at the first return 1 day visit and at 3 months after surgery
  Effectiveness of the pain control will be assessed by a 7-point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. Scale 1= Very much improved and scale 7 = very much worse
Satisfation of the pain control as per patients' report outcome | End of hospitalization (approximately 1 week after surgery)
  Enhance patient acceptance of the treatment by using oral administration, boosting confidence in the treatment plan and increasing adherence and effectiveness. Patient satisfaction and pain improvement will be assessed through a 5-point scale questionnaire. 1=very much discontent, 2=discontent, 3=fair, 4=satisfied, 5=very much satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Tsu-te Yeh, MD, Principal Investigator — TriService General Hospital
Locations (1):
- TriService General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Only anonymized and de-identified information can be collected from the participants as per institutional review board's approval.